CLINICAL TRIAL: NCT01808157
Title: A Phase II Randomised, Double Blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of CT327 Topical Ointment (0.05% and 0.5% w/w) Compared to Vehicle, in Subjects With Mild or Moderate Atopic Dermatitis and at Least Moderate Pruritus
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of CT327 in Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Creabilis SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT327-2005
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.05% w/w CT327 ointment (Experimental): Active
  Interventions: Drug: CT327 ointment
- 0.5% w/w CT327 ointment (Experimental): Active
  Interventions: Drug: CT327 ointment
- vehicle (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CT327 ointment
  Arms: 0.05% w/w CT327 ointment; 0.5% w/w CT327 ointment
Drug: placebo
  Arms: vehicle

SUMMARY:
This is a Phase II, multi-centre, randomised, double-blind, placebo-controlled study in male and female subjects, aged ≥ 12 years with mild/moderate atopic dermatitis and at least moderate pruritus. All subjects will receive BID topical applications of CT327 ointment or vehicle for up to 4 weeks.

At baseline, the subjects must have atopic dermatitis, as defined by the Hanifin and Rajka criteria, which involves a minimum of 5% and a maximum of 20% body surface area, an Investigator Global Assessment Score of 2 or 3 (mild or moderate) and pruritus visual analogue scale scores of ≥ 40mm (at least moderate).

All subjects will attend a screening visit not more than 21 days prior to Day 1. Subjects will be required to return to the clinic on Days 1 (baseline visit), 4, 11, 18 and 29 (end of treatment visit). All subjects will be asked to attend for a follow-up visit 14 (±3) days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects aged ≥ 12 years.

Clinical diagnosis of atopic dermatitis (as defined by Hanifin and Rajka criteria (Appendix F) at screening with:

* IGA score of 2 or 3 (mild or moderate)
* Score of ≥ 40mm on all screening pruritus VAS assessments (average and worst over the last 24 hours and current itch)
* A minimum of 5% and not more than 20% of the subjects' BSA affected by atopic dermatitis (affected is defined as active atopic dermatitis lesions or pruritus)
* Amenable to treatment with topical treatment
* Stable disease for ≥1 months prior to screening

Exclusion Criteria:

Atopic dermatitis only affecting the head or scalp. Unstable or actively infected atopic dermatitis. Concomitant dermatologic or medical condition(s) which may interfere with the investigator's ability to evaluate the subject's response to the study drug.

Subjects who have received monoclonal antibody therapy for their atopic dermatitis in the 4 months prior to screening.

Subjects who have used systemic immunosuppressive drugs, corticosteroids or received PUVA therapy in the 4 weeks prior to starting study treatment, or are scheduled to start these treatments during the study period.

Subjects who have used topical immunomodulators (pimecrolimus, tacrolimus) within 2 weeks of starting study treatment or are scheduled to start these treatments during the study period.

Subjects who have used topical corticosteroids from WHO group II, III or IV, or other treatments for atopic dermatitis, including wet wraps, within 2 weeks prior to starting study treatment or are likely to require treatment with these medications during the study period.

Subjects who are unable to abstain from using emollients from baseline (Visit 2) until the end of study treatment (Visit 6).

Subjects who are using any concomitant medication(s) that, in the investigators' opinion, could affect the subject's atopic dermatitis or pruritus (for example TADs, SSRI, pregabalin). Subjects using such medications may be included, at the investigators discretion, if they have been stable on treatment for at least 1 month prior to the start of study treatment and no changes to these medications are planned during the study period.

Subjects undergoing, or due to have, UVA, or UVB therapy in the 2 weeks prior to starting study treatment or during the study period.

Planned exposure of affected areas to excessive sunlight. Subjects with a clinically significant abnormal laboratory safety test and/or 12-lead ECG results at screening.

Subjects who are receiving any investigational drug or who have taken part in a clinical study with an investigational drug within three months prior to the start of study treatment.

Subjects with a known reaction or allergy to test drug or excipients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
• To determine whether CT327 is effective in reducing pruritus in subjects with atopic dermatitis, using a pruritus visual analogue scale (VAS) | 4 weeks

SECONDARY OUTCOMES:
• To assess efficacy of CT327 on atopic dermatitis using the Investigator Global Assessment (IGA) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Synexus, Manchester, Lancashire, Midlands, Wales, Scotland, United Kingdom